CLINICAL TRIAL: NCT00005477
Title: Hispanic and White Women's Cardiovascular Health
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4961; R03HL057100 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2002-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To elucidate the influence of ethnicity and socioeconomic status (SES) on women's cardiovascular health, using recently completed risk factor and mortality data from the Stanford Five-City Project.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

Two data sets were used to evaluate the specific aims: (1) survey risk factor data (e.g., blood pressure, cholesterol, blood lipids, smoking, etc.) on over 4500 girls and women; and (2) surveillance mortality data on over 1800 women.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-09; Study Completion 1998-08

REFERENCES:
- [Background] Behera SK, Winkleby MA, Collins R. Low awareness of cardiovascular disease risk among low-income African-American women. Am J Health Promot. 2000 May-Jun;14(5):301-5, iii. doi: 10.4278/0890-1171-14.5.301. PMID 11009856